CLINICAL TRIAL: NCT05565352
Title: Ketamine Treatment Safety and Tolerability in Psychiatric Inpatient Care Delivered at Depatment of Psychiatry, Medical University of Gdańsk, Poland
Brief Title: Ketamine Safety and Tolerability in Psychiatric Inpatient Care (KetGD)
Acronym: KetGD
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: NKBBN/172-447/2022
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder; Post Traumatic Stress Disorder; Obsessive-Compulsive Disorder; Somatoform Disorders; Anxiety Disorders; Dissociative Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder; Somatoform Disorders; Anxiety Disorders; Dissociative Disorders | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Major Depressive Disorder: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Major Depressive Disorder (MDD), as determined by a psychiatrist.
  Interventions: Drug: Ketamine Hydrochloride
- Obsessive Compulsive Disorder: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Obsessive Compulsive Disorder (OCD) as determined by a psychiatrist.
  Interventions: Drug: Ketamine Hydrochloride
- Post traumatic Stress Disorder: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Post-Traumatic Stress Disorder (PTSD) as determined by a psychiatrist.
  Interventions: Drug: Ketamine Hydrochloride
- Somatoform Disorder: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Somatoform Disorder as determined by a psychiatrist.
  Interventions: Drug: Ketamine Hydrochloride
- Anxiety Disorder: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Anxiety Disorder as determined by a psychiatrist.
  Interventions: Drug: Ketamine Hydrochloride
- Dissociative Disorder: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Dissociative Disorder as determined by a psychiatrist.
  Interventions: Drug: Ketamine Hydrochloride
- Bipolar Disorder: Patients must have a Diagnostic and Statistical Manual 5 (DSM-5) diagnosis of Bipolar Disorder as determined by a psychiatrist.
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine, a N-methyl-D-aspartate (NMDA) receptor antagonist has been used for general anesthesia since the 1970s, however, reports and trials by the end of the twentieth century and onward using subanesthetic doses suggested robust and rapid antidepressant and anti-suicidal effects. Ketamine is available as a 50/50 racemic mixture of enantiomers (S)-ketamine and (R)-ketamine.Ketamine will be infused (slow IV infusions of ketamine (0.5 mg/kg) over 40 minutes) twice weekly over a period of 4 weeks) Ketamine will be given in intranasal spray twice weekly over a period of 4 weeks Ketamine will be given orally (solution 2.0mg/kg, 2.5mg/kg) twice weekly over a period of 4 weeks.

SUMMARY:
This observational registry aims to collect real-world data on ketamine use in psychiatric inpatients within a regional tertiary-reference center. The study evaluates the safety and tolerability of ketamine administration in individuals with treatment-resistant mental disorders, characterized by diverse comorbidities, heterogeneous disease courses, and variations in treatment responses based on illness stage and severity with a subset of patients with remitted-recurrent and treatment-resistant or chronic presentations.

The registry is designed to systematically document adverse events, side effects, and patient-reported outcomes, providing a comprehensive assessment of both the short- and long-term effects of ketamine in psychopharmacology. By generating real-world evidence, this study shall contribute to a more nuanced understanding of ketamine's risk-benefit profile in clinical practice, particularly in subpopulations that are underrepresented in clinical trials. The findings prioritize the support for the refinement of treatment protocols and enhance patient safety in psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis as provided by DSM-5 criteria:

* Major depressive disorder (MDD),
* Bipolar disorder (BD),
* Anxiety disorder,
* Obsessive-compulsive disorder (OCD),
* Somatoform disorder,
* Post-traumatic stress disorder (PTSD),
* Dissociative disorder

Exclusion Criteria:

* Pregnancy and lactation
* Hypersensitivity to ketamine
* Uncontrolled hypertension
* Other uncontrolled somatic diseases that may impact safety per the investigator's judgment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients are referred to the tertiary-reference unit for mood disorders, anxiety disorders, obsessive-compulsive disorder, somatoform disorder, post-traumatic stress disorder, and dissociative disorder
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events assessed by Clinical-Administered Dissociative Symptoms Scale (CADSS) | Baseline through week 5
  Incidence of adverse events will be assessed by Clinician-Administered Dissociative Symptoms Scale (change from baseline to each measure). Higher values represent a worse severity, but not necessarily outcome. The Clinical-Administered Dissociative Symptoms Scale has 23-items based on dissociative symptoms during the assessment. Each item is scored 0 (normal) to 4 (severe symptoms) with overall score ranges from 0 (normal) to 92 (severe symptoms). Total number of assessments:18 times
Incidence of adverse events assessed by 4-items positive symptoms subscale of Brief Psychiatric Rating Scale (BPRS) | Baseline through week 5
  Incidence of adverse events will be assessed by 4-items positive symptoms subscale of Brief Psychiatric Rating Scale (change from baseline to each measure). Higher values represent a worse severity but not necessarily outcome. The 4-item positive symptoms subscale of Brief Psychiatric Rating Scale has 4-items based on conceptual disorganization, suspiciousness, hallucination and unusual thought content. Each item is scored 0 (normal) to 6 (severe symptoms) with overall score ranges from 0 (normal) to 24 (severe symptoms).
Incidence of adverse events assessed by body temperature (oral measurements) | Baseline through week 5
  Incidence of adverse events assessed by body temperature (oral measurement) in Celsius degree - change from baseline to each measure. A normal range is from 36.2 to 38.0 Celsius degrees; measurements beyond those ranges are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by blood pressure | Baseline through week 5
  Incidence of adverse events assessed by blood pressure (after the participant has rested for at least 5 minutes) in mmHg - change from baseline to each measure. A normal range for systolic blood pressure is from 90 to 140 mmHg, for diastolic blood pressure is from 50 to 90 mmHg; measurements beyond those ranges are clinically significant.
Incidence of adverse events assessed by respiration rate | Baseline through week 5
  Incidence of adverse events assessed by respiration rate in a breath number per minute - change from baseline to each measure. A normal range for respiration is from 12 to 16 breaths per minute; measurements beyond those ranges are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by pulse | Baseline through week 5
  Incidence of adverse events assessed by pulse (beats per minute [bpm]) - change from baseline to each measure. A normal range for pulse is from 60 to 90 bpm; measurements beyond those ranges are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by blood oxygen saturation | Baseline through week 5
  Incidence of adverse events assessed by blood oxygen saturation in percentage - change from baseline to each measure. A normal range for blood oxygen saturation is from 95 to 100 percentage; measurements under 95% are clinically significant. The total number of measurements: 44 times
Incidence of adverse events assessed by weight | Baseline through week 5
  Incidence of adverse events assessed by weight in kilograms- change from baseline to each measure. Gain weight for 7% baseline weight is clinically significant. Total numbers of assessments: 2. Weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Change in severity of depression symptoms assessed by Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline through week 5
  Change in severity of depression symptoms from baseline to each measure. Higher values represent a worse severity, but not necessarily outcome. The MADRS has 10-items which are based on mood symptoms over the past 7 days. Each item is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
Change in severity of symptoms assessed by Clinical Global Impression-Severity Scale (CGI-S) | Baseline through week 5
  CGI-S is a seven-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. CGI-S score starting from 1-not at all ending at 7-extremely severe.
Change in severity of symptoms assessed by Clinical Global Impression - Improvement Scale (CGI-I) | Baseline through week 5
  CGI-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.CGI-I score starting from 1-very much-improved ending at 7-very much worse
Change in severity of symptoms assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline through week 5
  C-SSRS is an assessment tool that evaluates suicidal ideation and behavior.
Change in severity of mania symptoms assessed by Young Mania Rating Scale (YMRS) | Baseline through week 5
  YMRS is an 11-item interviewer-rated scale used to evaluate manic symptoms at baseline and over time. The total scale score ranges from 0 to 60, where higher scores indicate more severe mania.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilkowska A, Wiglusz MS, Galuszko-Wegielnik M, Wlodarczyk A, Cubala WJ. Antianhedonic Effect of Repeated Ketamine Infusions in Patients With Treatment Resistant Depression. Front Psychiatry. 2021 Oct 18;12:704330. doi: 10.3389/fpsyt.2021.704330. eCollection 2021. PMID 34733182
- [Background] Wilkowska A, Wlodarczyk A, Galuszko-Wegielnik M, Wiglusz MS, Cubala WJ. Intravenous Ketamine Infusions in Treatment-Resistant Bipolar Depression: An Open-Label Naturalistic Observational Study. Neuropsychiatr Dis Treat. 2021 Aug 14;17:2637-2646. doi: 10.2147/NDT.S325000. eCollection 2021. PMID 34421299
- [Background] Wlodarczyk A, Cubala WJ, Galuszko-Wegielnik M, Szarmach J. Central nervous system-related safety and tolerability of add-on ketamine to antidepressant medication in treatment-resistant depression: focus on the unique safety profile of bipolar depression. Ther Adv Psychopharmacol. 2021 May 19;11:20451253211011021. doi: 10.1177/20451253211011021. eCollection 2021. PMID 34046159
- [Derived] Kachlik Z, Cubala WJ, Walaszek M, Pastuszak M, Pastuszak K, Kwasny A. Nonresponse to Ketamine in Treatment-Resistant Bipolar Depression. Neuropsychopharmacol Rep. 2025 Sep;45(3):e70038. doi: 10.1002/npr2.70038. PMID 40879542